CLINICAL TRIAL: NCT04885634
Title: Semaglutide for the Reduction of Arrhythmia Burden in Overweight and Obese Patients With Atrial Fibrillation (Pilot Study)
Brief Title: Semaglutide for the Reduction of Arrhythmia Burden in Overweight AF Patients
Acronym: SOCRATES-AF
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not received funding.
Sponsor: Axel Brandes (Other)
Collaborators: Herlev and Gentofte Hospital (Other); Hillerod Hospital, Denmark (Other); Svendborg Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Axel Brandes, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-SOCRATES-AF; 2021-002017-34 (EudraCT Number)
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation; Overweight and Obesity
Keywords: Atrial fibrillation; Overweight; Obesity; Semaglutide; Glucagon-like peptide-1 (GLP-1) receptor agonist; Implantable cardiac monitor
MeSH Terms: conditions — Atrial Fibrillation; Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Investigator-driven, prospective, parallel-group, double-blind, randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Semaglutide 2.4 mg subcutaneously once weekly in addition to standard AF care with lifestyle and risk factor management focusing on cardiovascular risk reduction
  Interventions: Drug: Semaglutide Injectable Product
- Control group (Placebo Comparator): Placebo treatment with volume-matched placebo s.c. once weekly in addition to standard AF care with lifestyle and risk factor management focusing on cardiovascular risk reduction
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Injectable Product — Subcutaneous injection of Semaglutide 2.4 mg once weekly
  Other Names: Semaglutide plus lifestyle and cardiovascular risk factor management
  Arms: Intervention group
Drug: Placebo — Subcutaneous injection of volume-matched placebo once weekly
  Other Names: Lifestyle and risk factor management alone
  Arms: Control group

SUMMARY:
The purpose of this pilot study is to assess the feasibility of a double-blind, randomized placebo-controlled trial of semaglutide 2.4 mg subcutaneously once weekly on top of standard care compared to standard care alone.

DETAILED DESCRIPTION:
The SOCRATES-AF pilot study is a prospective, parallel-group, double-blind, randomized controlled trial in patients with paroxysmal or early persistent atrial fibrillation and overweight and obesity.

The primary objective is to assess the feasibility of a double-blind, randomized placebo-controlled trial of semaglutide 2.4 mg subcutaneously (s.c.) once weekly on top of current standard care (lifestyle and risk factor management, oral anticoagulant and rate control therapy) versus current standard care alone in overweight or obese patients with symptomatic paroxysmal or early persistent AF.

To assess recurrences of atrial fibrillation all participants will receive an implantable cardiac monitor.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study-related activity
* ≥ 18 years of age at the time of signing informed consent
* Body mass index (BMI) ≥ 30 kg/m2
* Body mass index (BMI) ≥ 27 kg/m2 and at least 1 concomitant cardiometabolic risk factor (hypertension, dyslipidemia, or obstructive sleep apnea)
* Symptomatic paroxysmal or early persistent atrial fibrillation (Paroxysmal AF: Self- terminating, in most cases within 48 hours up to 7 days. AF episodes that are cardioverted within 7 days with a documented 12 lead ECG showing sinus rhythm within the last 12 months; early persistent AF: AF episodes lasting longer than 7 days, including episodes that are terminated by cardioversion, either with drugs or by direct current cardioversion, after 7 days or more. Early persistent AF in this trial is defined as persistent AF with first-time electrical cardioversion (ECV) or a maximum of 1 previous ECVs.)

Exclusion Criteria:

* General exclusion criteria

  * Age ≥75 years
  * History of type 1 or 2 diabetes (history of gestational diabetes is allowed)
  * Known or suspected hypersensitivity to study medication or related products
  * Treatment with GLP-1 receptor agonists within the last 3 months before randomisation
  * Treatment with dipeptidyl peptidase-4 (DPP-4) inhibitors
  * Alcohol/drug abuse
  * Pregnant or breastfeeding women
  * Fertile women not using chemical (tablet/pill, depot injection of progesterone, sub- dermal gestagen implantation, hormonal vaginal ring or transdermal hormonal patch) or mechanical (spirals) contraceptives
  * Active malignancy, unless in complete remission for ≥5 years
  * Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC)
  * Personal history of non-familial medullary thyroid carcinoma
  * Inflammatory bowel diseases
  * Acute or chronic pancreatitis
  * Obesity induced by other endocrinologic disorders (e.g. Cushing's Syndrome)
  * Current history of treatment with medications that may cause significant weight gain, within the last 3 months before screening, including systemic corticosteroids (except for a short course of treatment, i.e. 7-10 days), tri-cyclic antidepressants, atypical antipsychotic and mood stabilizers (e.g. imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid and its derivatives, and lithium)
  * Diet attempts using herbal supplements or over-the-counter medications within 3 months before screening
  * Current participation (or within the last 3 months) in an organised weight reduction programme or currently using or used within 3 months before screening: pramlintide, sibutramine, orlistat, zonisamide, topiramate, phentermine (either by prescription or as part of a clinical trial)
  * Severe chronic obstructive pulmonary disease
  * Uncontrolled treated/untreated hypertension (systolic >180 mmHg and/or diastolic >105 mmHg)
  * Previous or planned surgical treatment for obesity
  * Life expectancy <2.5 years
  * Other concomitant disease or treatment that according to the investigator's assessment makes the subject unsuitable for study participation
  * Participation in any other clinical intervention trial
  * Previous participation in the SOCRATES-AF pilot study
  * Inability to sign informed consent
* Exclusion criteria related to a cardiac condition

  * Previous or planned AF ablation
  * Previous use of continuous prophylactic class I or III antiarrhythmic drugs
  * Long-standing persistent or permanent AF
  * Overall clinical history of persistent AF ≥5 years
  * ECG suggestive of malignant ventricular arrhythmia
  * Prolonged corrected QT-interval (>500 ms), unless caused by bundle branch block
  * Myocardial infarction (MI) within the last 3 months before screening
  * Coronary revascularization within the last 3 months before screening
  * Planned coronary revascularisation
  * Cardiac surgery within the last 12 months before screening
  * Obstructive hypertrophic cardiomyopathy
  * Clinically significant valvular heart disease
  * Left ventricular (LV) dysfunction (HFrEF with left ventricular ejection fraction (LVEF) <45%) unless elicited by AF
  * Hospitalization due to decompensated heart disease within 30 days prior to randomization
  * Congestive heart failure (NYHA class IV)
  * Current myocardial or pericardial infection
  * Permanent pacemaker (PM) in use or implantable cardioverter defibrillator (ICD)
  * Patient cannot be prescribed non-vitamin K oral anticoagulant (NOAC)
  * perform physical exercise for medical or personal reasons
* Exclusion criteria based on laboratory abnormalities

  * Liver disease with increased plasma alanine aminotransferase (ALAT) levels of more than three times the upper limit of normal
  * Renal dysfunction (eGFR <30 ml/min), dialysis or kidney transplant
  * Clinically manifest thyroid dysfunction requiring therapy. After successful treatment of thyroid dysfunction, subjects may be enrolled, when thyroid function is controlled.
  * HbA1c >6.5% measured at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants to Complete Recruitment | Up to 68 weeks, until end of treatment
  Recruit 100 patients at an average recruitment rate of 2 patients per centre per month
Number of Participants to Complete Follow-up | Up to 75 weeks, until final follow-up
  Achieve complete follow-up on 90% or more of patients
Total Resource Requirement | Up to 75 weeks, until final follow-up
  Determine the resource requirements, i.e. primarily time spent per included patient, to achieve the recruitment and follow-up goals

SECONDARY OUTCOMES:
Efficacy of Semaglutide in Reducing AF Recurrences in Obese AF Patients | Up to 75 weeks, until final follow-up
  Collect preliminary information on the effect of semaglutide 2.4 mg s.c. once weekly on top of standard care on reducing AF recurrences in obese subjects with symptomatic paroxysmal or early persistent atrial fibrillation
Incidence of adverse effects of Semaglutide in overweight and obese AF patients | Up to 75 weeks, until final follow-up
  Collect preliminary information on adverse drug effects, which may lead to discontinuation or dose reduction

CONTACTS AND LOCATIONS:
Overall Officials: Axel Brandes, MD, DMSc, Study Director — Odense University Hospital; Morten L Hansen, MD, PhD, Study Director — Herlev and Gentofte Hospital

IPD SHARING:
Plan to Share IPD: No